CLINICAL TRIAL: NCT05043194
Title: The Preventive Study of Ursodeoxycholic Acid(UDCA) on Total Parenteral Nutrition Cholestasis(PNAC) in Premature Infants
Brief Title: Ursodeoxycholic Acid Prevents Total Parenteral Nutrition Cholestasis
Acronym: UDACPPNAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Liu (Other)
Responsible Party: Sponsor-Investigator, Wei Liu, Associate Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: wei liu
Record Dates: First submitted 2021-09-01; First posted 2021-09-14 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Cholestasis of Parenteral Nutrition
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ursodeoxycholic acid arm (Experimental): Premature infants who meet the inclusion criteria take preventive oral ursodeoxycholic acid on the 7th day after birth. ursodeoxycholic acid capsules (Ursofalk, 250 mg/capsules), starting with oral administration of pharmacologic doses of 20-25mg/kg/d, twice daily, until they were discharged .
  Interventions: Drug: Ursodeoxycholic Acid 250 Mg Oral Capsule
- the control arm (Sham Comparator): The control group was treated with UDCA after the occurrence of cholestasis.ursodeoxycholic acid capsules (Ursofalk, 250 mg/capsules), starting with oral administration of pharmacologic doses of 20-25mg/kg/d, twice daily, until they were discharged .
  Interventions: Drug: Ursodeoxycholic Acid 250 Mg Oral Capsule

INTERVENTIONS:
Drug: Ursodeoxycholic Acid 250 Mg Oral Capsule — prevention

SUMMARY:
This study aims to confirm whether the preventive use of ursodeoxycholic acid on the 5th day after birth in preterm infants who started parenteral nutrition therapy can reduce the occurrence of enteral nutrition-related cholestasis in preterm infants. This study examined the safety and efficacy of ursodeoxycholic acid (UDCA) in preventing Cholestasis Associated with Total Parenteral Nutrition in preterm infants.

DETAILED DESCRIPTION:
Investigators compared oral administration of UDCA prophylaxis with no prophylaxis in a randomized, open-label, proof-of-concept trial in preterm neonates with PN therapy.

ELIGIBILITY:
Inclusion Criteria:

1. admission to the hospital within 24 hours after birth
2. gestational ages:28-32 weeks
3. requiring TPN during the first days of life

Exclusion Criteria:

1. major congenital abnormalities, chromosomal abnormality congenital intrauterine infection, genetic metabolic diseases structural liver abnormality
2. surgical treatment was taken during hospitalization
3. with severe symptoms of digestive system disease before TPN
4. incompletion or withdrawal of treatment during hospitalization

Ages: 1 Day to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
direct bilirubin value of participants | up to 10 weeks
  Weekly direct bilirubin values in μmol/L for preterm infants during hospitalization will be collected to assess the severity of cholestasis

SECONDARY OUTCOMES:
The γ-GT activity level of participants | up to 10 weeks
  Weekly γ-GT values in U/L for preterm infants during hospitalization will be collected to assess the severity of cholestasis

CONTACTS AND LOCATIONS:
Overall Officials: liwen chang, Principal Investigator — Tongji Hospital
Locations (1):
- Wei Liu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No